CLINICAL TRIAL: NCT05494788
Title: Impact of CardiolRxTM on Recurrent Pericarditis An Open Label Pilot Study (MAvERIC-Pilot Study)
Brief Title: Impact of CardiolRxTM on Recurrent Pericarditis (MAvERIC-Pilot)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiol Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cardiol 100-004
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Pericarditis
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CardiolRx (Experimental): pharmaceutically produced Cannabidiol
  Interventions: Drug: CardiolRx

INTERVENTIONS:
Drug: CardiolRx — Oral solution
  Other Names: Pharmaceutically produced Cannabidiol

SUMMARY:
Patients with recurrent pericarditis who are refractory or intolerant to current therapeutic management options or who require long-term administration of corticosteroids to control their disease are particularly challenging to manage. The pathogenesis of pericarditis involves the activation of the inflammasome. CardiolRxTM (a pure cannabidiol [CBD] solution) is known to have anti-inflammatory properties, including modulation of inflammasome signaling. This pilot study is to assess the tolerance and safety of CardiolRxTM during the resolution of pericarditis symptoms, assess improvement in objective measures of disease, and during the extension period, assess the feasibility of weaning concomitant background therapy including corticosteroids while taking CardiolRxTM.

DETAILED DESCRIPTION:
Multi-center, open label Pilot Study. Patients who present with recurrent pericarditis will be screened and informed consent obtained.

Baseline assessments include the following: Clinical assessment, including vital signs, highest NRS pain score within the past 7 days of Day 1, 12-lead ECG; C-SSRS as well as hematology and blood chemistry and a pregnancy test for women with child-bearing potential.

Concomitant medications are recorded and any (S)AEs after informed consent has been obtained.

Study treatment will be initiated in the evening of Day 1, after all baseline assessments are completed.

Oral administration is as follows:

* Initial starting dose (Day 1 p.m. dose to Day 3 a.m. dose):

  5 mg/kg of body weight CardiolRxTM
* Day 3 p.m. dose to Day 10 a.m. dose: 7.5 mg/kg of body weight CardiolRxTM b.i.d.
* Day 10 p.m. dose to end of treatment period: 10.0 mg/kg of body weight CardiolRxTM b.i.d.

If the next higher dose after each study drug increase is not tolerated, the dose will be reduced to the previous tolerated dose.

Unless contraindicated in the opinion of the investigator, after 8 weeks of treatment, patients will enter an 18-week extension period (EP), in which they continue study treatment while their concomitant medications will be weaned.

Follow-up Procedures Every visit (before the next dose increase) the patient will be re-evaluated. This includes ECG monitoring at approximately 5 hours post-morning dose (Tmax) to surveil for deleterious effects on ECG intervals (particularly the QTc interval) and rhythm.

Drug titration will be dependent on investigator or designate interrogation of the ECGs and the absence of new, clinically significant abnormalities on those ECGs.

Vital signs, concurrent medication and (S)AEs will be recorded at all visits. Blood chemistry including liver function tests, hematology as well as INR assessments will be carried out at selected visits.

Final efficacy assessments will take place after 26 weeks of study treatment and include a clinical assessment, vital signs, pain score NRS, a 12-lead ECG, the C-SSRS, as well as laboratory assessments.

For patients who do not enter the EP, Final assessments will be done after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older
2. Diagnosis of at least two episodes of recurrent pericarditis*,
3. At least 1 day with pericarditis pain ≥4 on the 11-point Numerical Rating Scale (NRS) within prior 7 days
4. One of;

   1. C-Reactive Protein** (CRP) level ≥1.0 mg/dL within prior 7 days OR
   2. Evidence of pericardial inflammation assessed by delayed pericardial hyperenhancement on cardiac magnetic resonance imaging (CMR)
5. Currently receiving non-steroidal anti-inflammatory drugs (NSAIDs) and/or colchicine and/or corticosteroids (in any combination) for treatment of pericarditis in stable doses
6. Male patients with partners of childbearing potential who have had a vasectomy or are willing to use double barrier contraception methods during the conduct of the study and for 2 months after the last dose of study drug.
7. Women of childbearing potential willing to use an acceptable method of contraception starting with study drug administration and for a minimum of 2 months after study completion. Otherwise, women must be postmenopausal (at least 1 y absence of vaginal bleeding or spotting and confirmed by follicle stimulating hormone [FSH] ≥40 mIU/mL [or ≥ 40 IU/L] if less than 2 y postmenopausal) or be surgically sterile.

   * Diagnosis of pericarditis according to the 2015 European Society of Cardiology (ESC) Guidelines for the Diagnosis and Management of Pericardial Diseases (Adler et al. 2015):

At least two of:

1. Pericarditic chest pain
2. Pericardial rub
3. New widespread ST-segment elevation or PR-segment depression according to electrocardiogram (ECG) findings
4. Pericardial effusion (new or worsening)

   * Conversion: 1 mg/dL CRP = 10 mg/L hs-CRP

Exclusion Criteria:

1. Diagnosis of pericarditis that is secondary to specific prohibited etiologies, including tuberculosis (TB); neoplastic, purulent, or radiation etiologies; post-thoracic blunt trauma (e.g., motor vehicle accident); myocarditis
2. Estimated glomerular filtration rate (eGFR) <30 mL/min at screening
3. Elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 times the upper limit of normal (ULN) or ALT or AST >3x ULN plus bilirubin >2x ULN
4. Sepsis, defined as documented bacteremia at the time of screening or other documented active infection
5. Prior history of sustained ventricular arrhythmia
6. History of QT interval prolongation
7. QTc interval > 500 msec
8. Current participation in any research study involving investigational drugs or device
9. Inability or unwillingness to give informed consent
10. Ongoing drug or alcohol abuse
11. On any cannabinoid during the past month
12. Women who are pregnant or breastfeeding
13. Current diagnosis of cancer, with the exception of non-melanoma skin cancer
14. Any factor, which would make it unlikely that the patient can comply with the study procedures
15. Showing suicidal tendency as per the Columbia Suicide Severity Rating Scale (C-SSRS), administered at screening
16. On digoxin and/or type 1 or 3 antiarrhythmics
17. On immunosuppressive therapy with any of the following:

    1. Rilonacept
    2. Anakinra
    3. Canakinumab
    4. Methotrexate
    5. Azathioprine
    6. Cyclosporine
    7. Intravenous immune globulin (IVIG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen Klein, MD, Study Chair — The Cleveland Clinic
Locations (8):
- United States (8):
  - Pima Heart and Vascular Clinical Research, Tucson, Arizona
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University Health, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler Y, Charron P, Imazio M, Badano L, Baron-Esquivias G, Bogaert J, Brucato A, Gueret P, Klingel K, Lionis C, Maisch B, Mayosi B, Pavie A, Ristic AD, Sabate Tenas M, Seferovic P, Swedberg K, Tomkowski W; ESC Scientific Document Group. 2015 ESC Guidelines for the diagnosis and management of pericardial diseases: The Task Force for the Diagnosis and Management of Pericardial Diseases of the European Society of Cardiology (ESC)Endorsed by: The European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2015 Nov 7;36(42):2921-2964. doi: 10.1093/eurheartj/ehv318. Epub 2015 Aug 29. No abstract available. PMID 26320112
- [Background] Klein AL, Imazio M, Cremer P, Brucato A, Abbate A, Fang F, Insalaco A, LeWinter M, Lewis BS, Lin D, Luis SA, Nicholls SJ, Pano A, Wheeler A, Paolini JF; RHAPSODY Investigators. Phase 3 Trial of Interleukin-1 Trap Rilonacept in Recurrent Pericarditis. N Engl J Med. 2021 Jan 7;384(1):31-41. doi: 10.1056/NEJMoa2027892. Epub 2020 Nov 16. PMID 33200890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on January 9, 2023; Last patient last visit on September 6, 2024
Pre-assignment Details: 8-week follow up; 18-week extension period
Groups:
- CardiolRx: pharmaceutically produced Cannabidiol
  CardiolRx: Pharmaceutically produced Cannabidiol, titrated from 2.5/5 mg/kg of body weight to 10 mg/kg of body weight (or maximally tolerated dose), taken orally twice daily
Period: Initial Treatment Period
Arm/Group | CardiolRx
Started | 27
Completed | 24
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Period: Extension Period
Arm/Group | CardiolRx
Started | 24
Completed | 22
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- CardiolRx: pharmaceutically produced Cannabidiol
  CardiolRx: Pharmaceutically produced Cannabidiol
Arm/Group | CardiolRx
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (14.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
NRS Scores (Outcome measure 1) [Mean (Standard Deviation); unit: units on a scale] — Numerical Rating Scale for pain, patient self-reported within the past 7 days. Scale is from 0 to 10, with 0=no pain and 10=worst pain.
  units on a scale | 5.8 (1.71)
CRP [Mean (Standard Deviation); unit: mg/dl] | 4.44 (7.21)

OUTCOME MEASURES:

1. Primary Outcome: 11-point NRS Pain Score
Description: Change in pain score from baseline using 11-point NRS after 8 weeks of treatment. Nominal Rating Scale from 0 to 10, where 0 represents no pain and 10 maximum pain.
Time Frame: 8 weeks
Population: All patients enrolled
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CardiolRx
Number analyzed (Participants) | 27
units on a scale | -3.7 (2.07)

2. Other Pre Specified Outcome: Pericarditis Recurrence During the Extension Period (EP)
Description: Percentage of patients with pericarditis recurrence during the extension period (EP)
Time Frame: 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CardiolRx
Number analyzed (Participants) | 24
Participants | 7

3. Other Pre Specified Outcome: CRP Change From Baseline
Description: CRP change from baseline, as measured locally at baseline and at weeks 8, 16, and 26.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | CardiolRx
Number analyzed (Participants) | 22
mg/dl | 0.07 (0.10)

4. Other Pre Specified Outcome: Percentage of Patients With Normalized CRP Levels
Description: Percentage of patients with normalized CRP levels at 26 weeks (for patients with CRP ≥ 1.0 mg/dL at baseline)
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CardiolRx
Number analyzed (Participants) | 7
Participants | 7

5. Other Pre Specified Outcome: Percentage of Patients With Normalized CRP Levels
Description: Percentage of patients with normalized CRP levels at 8 weeks (for patients with CRP ≥1.0 mg/dL at baseline)
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | CardiolRx
Number analyzed (Participants) | 12
Participants | 7

6. Other Pre Specified Outcome: Time to Normalized CRP Levels
Description: Time to CRP normalization for patients with CRP ≥1.0 mg/dL at baseline
Time Frame: Over 26 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CardiolRx
Number analyzed (Participants) | 7
days | 26.4 (18.46)

7. Other Pre Specified Outcome: 11-point NRS Pain Score
Description: Change in pain score from baseline using 11-point NRS after 26 weeks of treatment. Nominal Rating Scale from 0 to 10, where 0 represents no pain and 10 maximum pain.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CardiolRx
Number analyzed (Participants) | 22
units on a scale | 4.3 (2.46)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signed ICF until the last study visit for each patient, up to 26 weeks.
Description: AE description does not differ from the clinical trials.gov AE definition.
  AEs were collected on an ongoing basis throughout the study.
Arm/Group | CardiolRx
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 1/27
Other Adverse Events (participants affected / at risk) | 14/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CardiolRx (N=27)
Chest pain (General disorders) | 1 (1)
ENTERITIS INFECTIOUS (Infections and infestations) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CardiolRx (N=27)
Pericarditis (Cardiac disorders) | 8 (10)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Chest discomfort (General disorders) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2)
INJURY, POISONING AND PROCEDURAL COMPLICATIONS (Injury, poisoning and procedural complications) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 7 (7)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 14 (14)
Nausea (Gastrointestinal disorders) | 5 (9)
Chest pain (General disorders) | 10 (13)
Fatigue (General disorders) | 5 (5)
Pain (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (7)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (2)
CRP increased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
In terms of limitations, this study was an open label, single-arm study so there was no control group. The number of patients included was also small but considered a sufficient sample size to demonstrate both the efficacy and safety objectives of this pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-01-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT05494788/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT05494788/SAP_001.pdf